CLINICAL TRIAL: NCT03990935
Title: Remineralization Potential of Ginger and Rosemary Herbals Versus Sodium Fluoride in Treatment of White Spot Lesions: "A Randomized Controlled Trial"
Brief Title: Remineralization Potential of Ginger and Rosemary Herbals Versus Sodium Fluoride in Treatment of White Spot Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nada Hamada Ahmed Shehab Eldin, resident at operative dentistry department,cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OPER - 607
Record Dates: First submitted 2019-06-13; First posted 2019-06-19 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: White Spot Lesions
MeSH Terms: interventions — ginger extract

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sodium fluoride varnish (Active Comparator): The fluoride varnish will be bifluorid 10 single use by voco (Germany). It Contains 5 % sodium fluoride (equal to 22,600 ppm fluoride).
  A thin coat will be applied on the tooth surface by using a brush. 10-20 s are sufficient for the varnish to be absorbed and then dry with air. Participants will be informed that they should not brush their teeth for 12-24 hours after the application and not to eat, or drink for at least 30 minutes after use to get the best results.
  Interventions: Other: ginger and rosemary gel
- Ginger and rosemary gel (Experimental): First the participant will be asked to brush his/her teeth thoroughly with 1450 ppm fluoride toothpaste (Colgate total healthy clean toothpaste). Then an application of a thin ribbon of this gel to the teeth using a brush. The medication will be left for at least 1 minute. The participant will be asked to spit out the medication after use and not to swallow it. Also the participant will be asked not to rinse his/her mouth, eat, or drink for at least 30 minutes after use to get the best results.
  Interventions: Other: ginger and rosemary gel

INTERVENTIONS:
Other: ginger and rosemary gel — First the participant will be asked to brush his/her teeth thoroughly with 1450 ppm fluoride toothpaste (Colgate total healthy clean toothpaste). Then an application of a thin ribbon of this gel to the teeth using a brush. The medication will be left for at least 1 minute. The participant will be asked to spit out the medication after use and not to swallow it. Also the participant will be asked not to rinse his/her mouth, eat, or drink for at least 30 minutes after use to get the best results.

SUMMARY:
To evaluate the effectiveness of ginger and rosemary herbals versus sodium fluoride in remineralization of incipient enamel caries.

DETAILED DESCRIPTION:
Group 1 (intervention)

Ginger and rosemary gel application:

First the participant will be asked to brush his/her teeth thoroughly with 1450 ppm fluoride toothpaste (Colgate total healthy clean toothpaste). Then an application of a thin ribbon of this gel to the teeth using a brush. The medication will be left for at least 1 minute. The participant will be asked to spit out the medication after use and not to swallow it. Also the participant will be asked not to rinse his/her mouth, eat, or drink for at least 30 minutes after use to get the best results.

Group 2 (control group). Sodium fluoride varnish The fluoride varnish will be bifluorid 10 single use by voco (Germany). It Contains 5 % sodium fluoride (equal to 22,600 ppm fluoride).

A thin coat will be applied on the tooth surface by using a brush. 10-20 s are sufficient for the varnish to be absorbed and then dry with air. Participants will be informed that they should not brush their teeth for 12-24 hours after the application and not to eat, or drink for at least 30 minutes after use to get the best results.

ELIGIBILITY:
Inclusion Criteria:

* Patient who has just completed a comprehensive orthodontic treatment.
* Presence of at least one WSL, DIAGNOdent score (0-20).
* Age range between 13 and 35years.

Exclusion Criteria:

* Patients with a compromised medical history.
* Severe or active periodontal disease
* Patients with developmental hypo-calcified lesions

Ages: 13 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-07 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
(white spot lesion progression) | T0 Baseline T1 1 months T2 3 months T3 6 months
  The change in the lesion fluorescence will be evaluated using diode laser fluorescence device (Diagnodent).

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt